CLINICAL TRIAL: NCT05193669
Title: VALidation of Tests Usable as a First Step TRIage to Manage Women Positive to High-risk Papillomavirus
Brief Title: Clinical Validation of Molecular Triage in HR-HPV Positive Women
Acronym: VALTRIHP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hiantis Srl (Industry)
Collaborators: European Commission (Other); Sciensano (Other Government); University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: WP7-HPVONC
Record Dates: First submitted 2021-12-11; First posted 2022-01-18 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cervical Carcinoma
Keywords: molecular HPV test; Pap-test; Triage
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Cervical swab, cervical biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Women accessing the HPV-based screening programme for primary screening, will undergo cervical sampling and clinical data recording. Samples from high-risk HPV positive women (around 2000 expected) will be aliquoted for testing with new HPV molecular test, that will allow full genotyping and viral load quantification.

ELIGIBILITY:
Inclusion Criteria:

* women participating in a cervical cancer screening program using an HPV assay as primary screening test
* positivity to hrHPV;
* written informed consent given.

Exclusion Criteria:

* total hysterectomy;
* diagnosis of CIN2+ in the last two years;
* hrHPV negative or inadequate.

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women accessing the HPV-based screening programme 'Prevenzione Serena', for primary screening, supported by a comprehensive follow-up registry.
Sampling Method: Non-Probability Sample
Enrollment: 23941 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the index triage test: Pap-test | Baseline
  Sensitivity of the index triage test(s) performed at the time of reflex testing for CIN2+ and CIN3+ detected at the time of reflex triage and relative sensitivity (index vs comparator)
Sensitivity of the index and comparator triage test: HPV molecular test | Baseline
  Sensitivity of the index and comparator triage test(s) performed at the time of reflex testing for CIN2+ and CIN3+ detected at the time of reflex triage + delayed triage; and relative sensitivity (index vs comparator).
Specificity of the index and comparator triage test | Month 12
  Specificity of the index and comparator triage test(s) performed at the time of reflex testing for <CIN2 considered at the time of reflex triage accepting negative colposcopy at the time of reflex testing and double negative index triage testing (reflex and delayed) as an acceptable proxy for <CIN2 and relative specificity for <CIN2 (index vs comparator).

CONTACTS AND LOCATIONS:
Overall Officials: Paola Armaroli, MD, Principal Investigator — AOU Città della Salute e della Scienza di Torino, Itay; Marc Arbyn, MD, Study Director — Sciensano - Brussels, Belgium
Locations (1):
- AOU Città della Salute e della Scienza di Torino S.S.D. Epidemiologia, Screening- CPO, Torino, Italy